CLINICAL TRIAL: NCT03710044
Title: Investigation of Flare and Remission in Atopic Dermatitis in an Integrated Longitudinal Trial: Effects of Systemic Treatment With Cyclosporine A
Brief Title: Investigation of Flare and Remission in Subjects With Atopic Dermatitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EXP-1392; 2018-000229-30 (EudraCT Number)
Record Dates: First submitted 2018-10-16; First posted 2018-10-17 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2019-07

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; cyclosporine A; atopic dermatitis pathophysiology
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclosporine A treatment (Experimental): Oral cyclosporine A treatment
  Interventions: Drug: Cyclosporine A

INTERVENTIONS:
Drug: Cyclosporine A — Initial treatment: Oral cyclosporine A (CsA) treatment (4-5 mg/kg/day) for 3 weeks.
  Responders shift to oral low-dose CsA treatment (2-2.5 mg/kg/day) until onset of a second flare or until Week 16 (Day 113).
  In case of a second AD flare, the subjects shift back to oral high-dose CsA treatment (4-5 mg/kg/day) for 3 weeks.

SUMMARY:
The trial is an exploratory, single-centre, uncontrolled, open-label, interventional trial of up to 19 weeks' duration to investigate flare and remission in subjects with moderate-to-severe atopic dermatitis (AD) treated with cyclosporine A (CsA).

DETAILED DESCRIPTION:
40 subjects with moderate-to-severe AD will be treated with a 3-week course of high-dose CsA, which is a standard-of-care treatment regimen. After 3 weeks, all responders shift to oral low-dose CsA treatment (2-2.5 mg/kg/day) until onset of a second flare or until Week 16 (Day 113).

In case of a second AD flare, the subjects shift back to oral high-dose CsA treatment (4-5 mg/kg/day) for 3 weeks.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis and history of chronic, moderate-to-severe AD (by the Eichenfield revised criteria of Hanifin and Rajka) for at least 3 years before the screening visit.
* Subjects who have an AD flare at the start of the trial (EASI score ≥10 at screening and ≥16 at the baseline visit).

Main Exclusion Criteria:

* Treatment with allergen immunotherapy within 6 months before the baseline visit.
* Treatment with leukotriene inhibitors, systemic glucocorticoids, or other systemic treatment for AD (including immunosuppressive treatment, ultraviolet therapy, and biologics) within 4 weeks before the baseline visit.
* Treatment with topical corticosteroids or topical calcineurin inhibitors within 1 week before the baseline visit.
* Chronic or acute infection requiring treatment with oral or intravenous antibiotics, anti-virals, anti-parasitics, anti-protozoals, or anti-fungals within 4 weeks before the screening visit or superficial skin infections within 1 week before the screening visit.
* History of malignancy within 5 years before the baseline visit, with the following exceptions: subjects with a history of completely treated carcinoma in situ of cervix, and non-metastatic squamous or basal cell carcinoma of the skin are allowed.
* Hypertension (>150/95 mmHg) at the screening visit.
* Planned surgical procedure during the length of the subject's participation in this trial.
* Use of a tanning booth/parlour within 4 weeks before the screening visit.
* Pregnant, breastfeeding, or lactating women.
* Laboratory abnormalities at the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Time to flare* in subjects with moderate-to-severe AD who responded to a 3-week course of high-dose CsA treatment. | Day 1 to Day 113 (end of trial)
  *A flare is defined as exacerbation of the disease, where intensification of medicine is considered necessary.

SECONDARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) up until end of trial. | Up to Day 113 (end of trial)
Number of subjects with TEAEs up until end of trial. | Up to Day 113 (end of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- Investigational site, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No